CLINICAL TRIAL: NCT02363738
Title: A Multisite, Fixed Dose, Randomized, Double-Blind, Placebo-Controlled 12-Week Study Evaluating the Efficacy, Safety, and Tolerability of Adjunctive Infliximab for the Treatment of Bipolar I/II Depression
Brief Title: 12-Week Study Evaluating the Efficacy, Safety, and Tolerability of Adjunctive Infliximab for Bipolar I/II Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Infliximab-BD
Record Dates: First submitted 2015-01-05; First posted 2015-02-16 (Estimated); Results first posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-06

CONDITIONS: Bipolar Depression
Keywords: Bipolar Disorder; Bipolar Depression; Inflammation; Bipolar
MeSH Terms: conditions — Bipolar Disorder; Inflammation | interventions — Infliximab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infliximab (Experimental): Intravenous infliximab (5mg/kg) at baseline, week 2 and 6 under clinical observation
  Interventions: Drug: Infliximab
- Saline (Placebo) (Placebo Comparator): Intravenous placebo (saline solution) at baseline, week 2 and 6 under clinical observation. Placebo will be matched to infliximab in color and consistency.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Infliximab — Intravenous infliximab (5mg/kg) at baseline, week 2 and 6 under clinical observation. Infliximab will be prescribed adjunctively to a conventional mood stabilizer or atypical antipsychotic agent.
  Other Names: Remicade
  Arms: Infliximab
Other: Saline — Intravenous placebo (saline solution) at baseline, week 2 and 6 under clinical observation. Placebo will be matched to infliximab in color and consistency and will be administered adjunctively to conventional mood stabilizer or atypical antipsychotic agent.
  Arms: Saline (Placebo)

SUMMARY:
Studies show the presence of immuno-inflammatory disturbances in individuals with Bipolar Disorders (BD). Increased levels of circulating proteins known as cytokines that promote inflammation have been consistently reported in individuals with bipolar disorders. A particular cytokine referred to as Tumor Necrosis Factor (TNF)-alpha is among those cytokines that have been consistently identified across depressive, manic, and euthymic periods. Disturbances in inflammation however, are not seen in all individual with bipolar disorder. Those individuals with signs of inflammation also often present with higher prevalence of medical disorders that are also associated with inflammation. Those individuals with significant signs of inflammation may respond to anti-inflammatory treatments. In this study, individuals with bipolar depression who exhibit signs of high inflammation will be enrolled and treated with either an anti-inflammatory biologic known as infliximab or placebo (saline).

ELIGIBILITY:
Inclusion Criteria:

* Fifth edition of Diagnostic and Statistical Manual for Mental Disorders (DSM-5) criteria for major depressive episode as part of bipolar I/II disorder and are able to provide written informed consent
* HAMD-17 score >= 20
* Young Mania Rating Scale score < 12
* Previous failed trial (i.e., inefficacy) of quetiapine and one other Canadian Network for Mood and Anxiety Treatments (CANMAT) BD guideline/FDA approved first line treatment for the depressive phase of BD during the index episode and/or during a prior episode
* Currently prescribed conventional mood stabilizer or atypical antipsychotic agent
* Received conventional treatment for bipolar depression for a minimum of 4 weeks prior to randomization
* Females of childbearing potential must test negative for pregnancy and must be using adequate birth control measures throughout the study and must continue such precautions for 6 months after receiving the last study drug administration.

Participants will also need to meet one of the following inflammatory indicators:

1. Central Obesity (ethnicity-specific waist circumference - see table below for specific values) OR BMI ≥30 kg/m2.

   AND
   * Raised triglycerides: ≥1.7 mmol/L (150 mg/dL) or specific treatment for this lipid abnormality OR
   * Reduced HDL-cholesterol: <1.03 mmol/L (40 mg/dL) in males; <1.29 mmol/L (50 mg/dL) in females or specific treatment for this lipid abnormality OR
   * Raised Blood Pressure: Raised blood pressure Systolic: ≥130 mm Hg or diastolic: ≥85 mm Hg or treatment of previously diagnosed hypertension.
2. Diabetes: 8-hour fasting plasma glucose ≥ 7.0 mmol/L or Hb-A1C test ≥ 6.5% (as per the 2013 CDA diagnostic criteria) or previously diagnosed type 1 or 2 diabetes (current prescription medication for diabetes acceptable of diagnosis). Participants with child onset of diabetes will be excluded.
3. Inflammatory bowel disorder (Ulcerative Colitis, Crohn's disease).
4. Rheumatological disorders (rheumatoid arthiristis); Psoriasis.
5. Smoking cigarettes (daily - minimum of ½ pack).
6. High sensitivity C-reactive protein level of ≥5 mg/L via blood test at screening

Exclusion Criteria:

* Another concurrent psychiatric disorder that requires primary clinical attention
* History of schizophrenia
* Active psychotic symptoms
* Substance abuse and/or dependence within past 6 months
* Electroconvulsive therapy in the past 6 months
* Actively suicidal or evaluated as being a suicide risk [HAMD-17 suicide item >= 3 or Montogomery Asberg Depression Rating Scale (MADRS) suicide item >= 4, or according to clinical judgement using the C-SSRS]
* Clinically significant unstable medical illness
* Severe infections such as sepsis, abscess, tuberculosis and opportunistic infections
* Viral hepatitis B
* History of Hepatitis C ( documented or suspected)
* Any autoimmune disorder
* History of tuberculosis or a high risk of tuberculosis exposure
* Human Immunodeficiency Virus confirmed by laboratory testing
* Active fungal infection
* History of recurrent viral or bacterial infections
* Received within 3 months prior to screening or are expected to receive any live viral vaccine or live bacterial vaccinations during the trial or up to 3 months after the last administration of study agent
* C. difficile infection within the past 4 months
* History of lymphoproliferative disease
* History of cancer, excluding basal cell or squamous cell carcinoma of the skin (fully excised with no recurrence)
* Unstable cardiovascular, endocrinological, hematological, hepatic, renal or neurological disease determined by physical examination and laboratory testing
* Concomitant diagnosis or any history of congestive heart failure
* Concomitant treatment with non-steroidal and steroidal anti-inflammatory medications or other biologics
* Current or past exposure to anti-TNF biologics
* Previous immediate hypersensitivity response, including anaphylaxis to an immunoglobulin product (plasma-derived or recombinant, e.g. monoclonal antibody)
* Known allergies, hypersensitivity or intolerance to infliximab or its excipients
* Known allergy to murine proteins or other chimeric proteins
* Currently on or have used any investigational drug within 30 days prior to screening, or within 5 half-lives of the investigational agent
* Females who are pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger S McIntyre, MD, FRCPC, Principal Investigator — University of Toronto; University Health Network
Locations (2):
- VA Palo Alto Health Care System, Palo Alto, California, United States
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lee Y, Mansur RB, Brietzke E, Carmona NE, Subramaniapillai M, Pan Z, Shekotikhina M, Rosenblat JD, Suppes T, Cosgrove VE, Kramer NE, McIntyre RS. Efficacy of adjunctive infliximab vs. placebo in the treatment of anhedonia in bipolar I/II depression. Brain Behav Immun. 2020 Aug;88:631-639. doi: 10.1016/j.bbi.2020.04.063. Epub 2020 May 4. PMID 32380271
- [Derived] McIntyre RS, Subramaniapillai M, Lee Y, Pan Z, Carmona NE, Shekotikhina M, Rosenblat JD, Brietzke E, Soczynska JK, Cosgrove VE, Miller S, Fischer EG, Kramer NE, Dunlap K, Suppes T, Mansur RB. Efficacy of Adjunctive Infliximab vs Placebo in the Treatment of Adults With Bipolar I/II Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Aug 1;76(8):783-790. doi: 10.1001/jamapsychiatry.2019.0779. PMID 31066887
- [Derived] Lee Y, Subramaniapillai M, Brietzke E, Mansur RB, Ho RC, Yim SJ, McIntyre RS. Anti-cytokine agents for anhedonia: targeting inflammation and the immune system to treat dimensional disturbances in depression. Ther Adv Psychopharmacol. 2018 Nov 19;8(12):337-348. doi: 10.1177/2045125318791944. eCollection 2018 Dec. PMID 30524702

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infliximab | Saline (Placebo)
Started | 29 | 31
Completed | 21 | 26
Not Completed | 8 | 5
Not completed — Adverse Event | 5 | 2
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: One participant was excluded from the Infliximab arm and 1 participant was excluded from placebo arm of the study because they did not complete at least 1 efficacy assessment after baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Infliximab | Saline (Placebo) | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (11.7) | 46.8 (10.2) | 45.71 (10.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 26 | 46
  Male | 8 | 4 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 24 | 48
  Other | 4 | 6 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 26 | 27 | 53
  United States | 2 | 3 | 5
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.5 (10) | 34.6 (8) | 34.5 (8.95)
Number of lifetime psychiatric hospitalizations [Mean (Standard Deviation); unit: Hospitalizations] | 1.8 (1.9) | 1.6 (2.0) | 1.65 (2.0)
Baseline MADRS total score [Mean (Standard Deviation); unit: units on a scale] — The baseline Montgomery-Asberg Depression Rating Scale (MADRS) score is used to assess the baseline depressive symptoms. The range of possible values on the scale is 0 to 60. The higher the score, the worse the overall depressive symptoms.
  units on a scale | 30.6 (7.2) | 29.5 (7) | 30 (7.01)
Baseline YMRS total score [Mean (Standard Deviation); unit: units on a scale] — The Young Mania Rating Scale (YMRS) total score ranges from 0 to 60, where higher scores indicate more severe mania.
  units on a scale | 3.5 (3.0) | 4.4 (4.2) | 3.9 (3.5)
Bipolar I disorder [Count of Participants; unit: Participants] | 16 | 15 | 31
Bipolar II disorder [Count of Participants; unit: Participants] | 12 | 15 | 27
Educational level [Count of Participants; unit: Participants]
  High school | 6 | 5 | 11
  College or university | 17 | 24 | 41
  Graduate school | 5 | 1 | 6
CRP level, age-adjusted [Mean (Standard Deviation); unit: mg/L] | 4.5 (3.3) | 7.3 (8.1) | 7.0 (8.3)
Inflammatory criteria met [Count of Participants; unit: Participants]
  CRP level greater than or equal to 5 mg/L | 10 | 15 | 25
  Obesity combined with hypertension or dyslipidemia | 20 | 25 | 45
  Diabetes type 1 or 2 | 7 | 5 | 12
  Inflammatory bowel disorder | 1 | 2 | 3
  Rheumatologic disorder | 6 | 8 | 14
  Daily cigarette smoking | 6 | 8 | 14
  Migraine headaches | 9 | 7 | 16
Medications [Count of Participants; unit: Participants]
  Lithium carbonate | 6 | 5 | 11
  Valproate sodium | 5 | 3 | 8
  Quetiapine fumarate | 8 | 5 | 13
  Olanzapine and fluoxetine hydrochloride | 0 | 1 | 1
  Lurasidone hydrochloride | 4 | 5 | 9
  Lamotrigine | 8 | 7 | 15
  Antidepressant | 13 | 20 | 33

OUTCOME MEASURES:

1. Primary Outcome: Baseline and Week 12 Montgomery-Asberg Depression Rating Scale (MADRS) Scores
Description: Baseline and Week 12 Montgomery-Asberg Depression Rating Scale scores are provided, with the range of possible values on the scale from 0 to 60. The higher the score, the worse the overall depressive symptoms.
Time Frame: Up to 12 weeks
Population: The modified intent-to-treat analysis included all participants who had received at least 1 infusion of study medication and completed at least 1 after-baseline efficacy assessment. One participant from the Infliximab arm and one participant from the placebo arm were excluded fromt he analyses because they did not complete at least one efficacy assessment after baseline.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Infliximab | Saline (Placebo)
Number analyzed (Participants) | 28 | 30
units on a scale
  Baseline | 29.61 (1.36) | 27.79 (1.59)
  Week. 12 | 18.64 (2.40) | 16.06 (2.00)

2. Primary Outcome: Baseline and Week 6 Montgomery-Asberg Depression Rating Scale (MADRS) Scores
Description: Baseline and Week 6 Montgomery-Asberg Depression Rating Scale (MADRS) scores, where the range of possible values on the scale is from 0 to 60. The higher the score, the worse the overall depressive symptoms.
Time Frame: Up to 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Infliximab | Saline (Placebo)
Number analyzed (Participants) | 28 | 30
units on a scale
  Baseline | 29.61 (1.36) | 27.79 (1.59)
  Week 6 | 19.44 (2.27) | 20.94 (2.29)

3. Secondary Outcome: Changes in Brain N-acetylaspartate Levels
Description: Changes in prefrontal metabolites concentration of N-acetylaspartate, using proton-magnetic resonance spectroscopy (1H-MRS), adjusted for age, sex, baseline values and % gray matter in the spectroscopic region of interest.
Time Frame: Baseline to Week 12
Population: The number of total participants analyzed is lower than those previously reported in the primary outcome measure as only a subgroup of participants underwent this additional and optional MRS testing.
Measure: Least Squares Mean (Standard Error); unit: mmol/kg
Arm/Group | Infliximab | Saline (Placebo)
Number analyzed (Participants) | 15 | 18
mmol/kg
  Baseline | 5.67 (0.09) | 5.65 (0.09)
  Week 12 | 5.71 (0.21) | 5.81 (0.18)

4. Secondary Outcome: Changes in Anhedonia
Description: Change in the Snaith-Hamilton Pleasure Scale (SHAPS) total score. Total score range of 14 to 56, with greater scores indicative of greater hedonic capacity.
Time Frame: Baseline to 12 weeks
Population: Three participants in the Infliximab group did not complete at least one post-baseline efficacy assessment. Three participants did not complete at least one post-baseline efficacy assessment.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Infliximab | Saline (Placebo)
Number analyzed (Participants) | 25 | 27
Score on a scale
  Baseline | 34.04 (1.73) | 34.8 (1.45)
  Week 12: number analyzed (Participants) | 21 | 26
  Week 12 | 37.17 (1.5) | 40.79 (1.69)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from screening (prior to baseline) through the completion of the study at week 12 (minimum of 3 months).
Arm/Group | Infliximab | Saline (Placebo)
All-Cause Mortality (participants affected / at risk) | 1/29 | 1/31
Serious Adverse Events (participants affected / at risk) | 1/29 | 2/31
Other Adverse Events (participants affected / at risk) | 4/29 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=29) | Saline (Placebo) (N=31)
Mortality (Nervous system disorders) | 1 (1) | 0 (0) — A participant who received infliximab at the Stanford site died due to anoxic brain injury approximately 4 weeks after the third infusion.
Mortality (Social circumstances) | 0 (0) | 1 (1)
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3.44% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=29) | Saline (Placebo) (N=31)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hair loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Reactive arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abnormal liver function enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0) — Replicated abnormalities in laboratory assessments of liver function (ie, alanine aminotransferase and aspartate aminotransferase levels) without associated symptoms after 2 infusions of infliximab, patient dismissed from study before third infusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT02363738/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT02363738/ICF_001.pdf